CLINICAL TRIAL: NCT05795543
Title: Single Versus Double Screws Fixation of Subtalar Arthrodesis : A Prospective Randomized Controlled Study
Brief Title: Subtalar Arthrodesis by Single Versus Double Screws
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mahmoud moustafa khalafallah ali, Qena, Eygpt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: subtalar arthrodesis
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Subtalar Osteoarthritis Secondary to Inflammatory Arthritis
Keywords: subtalar arthrodesis; screws

STUDY DESIGN:
Intervention Model Description: participant divide to 2 groups first group subtalar arthrodesis by single screw second group subtalar arthrodesis by double screws
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): subtalar arthrodesis by single screw
  Interventions: Procedure: Subtalar Arthrodesis by Screws
- B (Active Comparator): subtalar arthrodesis by double screws
  Interventions: Procedure: Subtalar Arthrodesis by Screws

INTERVENTIONS:
Procedure: Subtalar Arthrodesis by Screws — Instruments: cannulated screws Steps: supine position , tournique over the thigh, using a extended lateral approach or sinus tarsi approach with joint debridement and preparation. Single-screw fixation was most often placed from posterior to anterior and double screws fixation was placed triangular pattern

SUMMARY:
Compare clinical and radiological outcome of use of single screw versus double screws fixation for subtalar arthrodesis

DETAILED DESCRIPTION:
The subtalar joint consists of an anterior, posterior and medial joint facet, which allows for inversion - and eversion of the foot. Several pathologies may lead to pain originating from the subtalar joint, including primary arthritis, posttraumatic arthritis, congenital or acquired deformities, instability, tarsal coalition or inflammatory diseases Management of these pathologies variable including conservative and operative treatment once conservative treatment has failed subtalar fusion is a common surgical procedure which is a well-established and widely accepted There are many surgical techniques described for fusion , one of these techniques is fixation with screws The rate of non-union varies among authors between 0-46%, that's may due to lack of standardization of techniques should be used

ELIGIBILITY:
Inclusion Criteria:

* All patients who will be operated by subtalar fusion for any indication Age range 18 - 65

Exclusion Criteria:

* Age < 18 years , > 65 Acute calceneal fracture Infection Non union Bone defect that need bone graft Refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fusion rate | 3 month
  subtalar fusion radiologically and clinically

SECONDARY OUTCOMES:
Functional assessment -rate of complications(e.g. non-union, post-operative infections, Instability) -secondary surgery procedures | 3 month
  by AOFAS Ankle-Hindfoot Scale

REFERENCES:
- [Background] Wirth SH, Viehofer A, Fritz Y, Zimmermann SM, Rigling D, Urbanschitz L. How many screws are necessary for subtalar fusion? A retrospective study. Foot Ankle Surg. 2020 Aug;26(6):699-702. doi: 10.1016/j.fas.2019.08.017. Epub 2019 Sep 6. PMID 31522872
- [Background] Buch BD, Myerson MS, Miller SD. Primary subtaler arthrodesis for the treatment of comminuted calcaneal fractures. Foot Ankle Int. 1996 Feb;17(2):61-70. doi: 10.1177/107110079601700202. PMID 8919403